CLINICAL TRIAL: NCT06996353
Title: Clinical Data Collection of Myopic Patients After PTK-PRK With CZM MEL 90 Excimer Laser for Verification of Predicted Refractive Outcome Using EpiMaster Software Considering Epithelial Remodelling
Brief Title: Clinical Data Collection of Myopic Patients After PTK-PRK With CZM MEL 90 Excimer Laser
Status: Recruiting | Type: Observational
Sponsor: London Vision Clinic (Other)
Collaborators: Optana GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: LoVC-011
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PTK-PRK refractive treatment — The PTK-PRK refractive treatment will be done according to routine clinical practice.

SUMMARY:
The objective of the clinical investigation presented to is to verify predictions of post-operative PTK-PRK refractive outcome made by the EpiMaster application software by comparing these to post-operative clinical data after routine PTK-PRK treatments.

DETAILED DESCRIPTION:
The objective of the clinical investigation presented to is to verify predictions of post-operative PTK-PRK refractive outcome made by the EpiMaster application software by comparing these to post-operative clinical data after routine PTK-PRK treatments.

The EpiMaster application software is not used in this clinical investigation, consequently, it is a merely observational investigation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are according to the user manual of CZM MEL 90 Excimer Laser for treatment of refractive errors
* Patient present with myopic or myopic and astigmatic error
* Patient will be able to understand the patient information and willing to sign an informed consent
* Patient will be willing to comply with all follow-up visits and the respective examinations

Exclusion Criteria:

* Exclusion criteria are according to the user manual of CZM MEL 90 Excimer Laser for treatment of refractive errors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient present with myopic or myopic and astigmatic error
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Difference of SE(measured) and SE(predicted by EpiMaster) | 6 months
  Percentage of eyes with SE6 months post-op "measured" - SEpredicted by EpiMaster within ±1.00D, with SE being the spherical equivalent

CONTACTS AND LOCATIONS:
Overall Officials: Dan Z Reinstein, MD, Study Director — London Vision Clinic Ltd., London, United Kingdom; Sheetal Brar, MD, Principal Investigator — Pro Sight Eye Hospital, Chandigarh, India; Aadithreya Varman, MD, Principal Investigator — Uma Eye Clinic, Chennai, India
Locations (2):
- India (2):
  - Pro Sight Eye Hospital, Chandigarh, Punjab Haryana
  - Uma Eye Clinic, Chennai, Tamil Nadu

IPD SHARING:
Plan to Share IPD: No
The plan is to not share IPD.